CLINICAL TRIAL: NCT03914443
Title: A Feasibility Trial of Nivolumab With Neoadjuvant CF or DCF Therapy for Locally Advanced Esophageal Carcinoma FRONTiER Trial
Brief Title: A Feasibility Trial of Nivolumab With Neoadjuvant CF or DCF Therapy for Locally Advanced Esophageal Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Center, Japan (Other Government)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry); Fiverings Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JCOG1804E
Record Dates: First submitted 2019-04-11; First posted 2019-04-16 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Locally Advanced Esophageal Squamous Cell Carcinoma
Keywords: Esophageal squamous cell carcinoma; Neoadjuvant chemotherapy; Nivolumab; JCOG
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Nivolumab; Fluorouracil; Cisplatin; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cohort A (Experimental): "Nivolumab: 360 mg, every 3 week 5-FU: 800 mg/m^2, every 3 week CDDP: 80 mg/m^2, every 3 week "
  Interventions: Biological: Nivolumab; Drug: 5-FU; Drug: CDDP
- Cohort B (Experimental): "Nivolumab: 240 mg lead-in followed by 360 mg, every 3 week 5-FU: 800 mg/m^2, every 3 week CDDP: 80 mg/m^2, every 3 week "
  Interventions: Biological: Nivolumab; Drug: 5-FU; Drug: CDDP
- Cohort C (Experimental): "Nivolumab: 360 mg, every 3 week 5-FU: 750 mg/m^2, every 3 week CDDP: 70 mg/m^2, every 3 week DTX: 70mg/m^2, every 3 weeks"
  Interventions: Biological: Nivolumab; Drug: 5-FU; Drug: CDDP; Drug: DTX
- Cohort D (Experimental): "Nivolumab: 240 mg lead-in followed by 360 mg, every 3 week 5-FU: 750 mg/m^2, every 3 week CDDP: 70 mg/m^2, every 3 week DTX: 70mg/m^2, every 3 weeks"
  Interventions: Biological: Nivolumab; Drug: 5-FU; Drug: CDDP; Drug: DTX

INTERVENTIONS:
Biological: Nivolumab — 240 mg or 360 mg
  Other Names: ONO-4538
Drug: 5-FU — 750 or 800 mg^2
  Other Names: 5-Fluorouracil
Drug: CDDP — 70 or 80 mg/m^2
  Other Names: Cisplatin
Drug: DTX — 70 mg/m^2
  Other Names: Docetaxel
  Arms: Cohort C; Cohort D

SUMMARY:
The main purpose of this study is to evaluate the safety of the neoadjuvant therapy, nivolumab with CF (5-FU, CDDP) or nivolumab with DCF (5-FU, CDDP, DTX), for locally advanced esophageal carcinoma.

ELIGIBILITY:
Inclusion criteria:

1. Endoscopic biopsy of esophageal primary lesion histologically diagnosed as squamous cell carcinoma, adenosquamous carcinoma, or basal cell carcinoma
2. All esophageal cancer lesions are localized in the thoracic esophagus
3. Patients are classified as clinical stage T1N1-3M0 or T2-3N0-3M0 in the UICC-TNM classification 8th edition
4. The age is over 20 years old and under 75 on the enrollment date
5. PS 0-1
6. With or without measurable lesions
7. Patients who have no medical history of treatment for esophageal cancer
8. Patients who have no medical history of chemotherapy, radiotherapy, and endocrine therapy, including treatment for other types of cancer
9. The results of laboratory tests within 14 days before enrollment meet the inclusion criteria
10. Esophageal cancer radical surgery (R0) by open-chest surgery (or thoracoscopic surgery) and laparotomy (or laparoscopic surgery) is judged possible
11. Patients who have no complication or history of thyroid dysfunction
12. Patients who have no complication or history of autoimmune disease
13. Patients who don't have treatment with systemic corticosteroids (dose of 10mg/day over in prednisolone equivalent) or immunosuppressants within 14 days before enrollment
14. Patients who have no complication or history of pneumonitis or pulmonary fibrosis which had been diagnosed by imaging tests or physical examination
15. For females, who have agreed with contraception from start of investigational drug administration to 5 months after last dose of an investigational drug. For males who have agreed with contraception from start of investigational drug administration to 7 months after last dose of an investigational drug.
16. Obtained written informed consent from patients"

Exclusion criteria:

1. Patients who have active multiple cancers
2. Patients who have an infectious disease that is active and need the systemic treatment
3. Positive with HBs antigen, HCV-RNA or anti-HIV antibody, or anti-HTLV-1 antibody tests
4. Negative with HBs antigen test and positive with anti HBs antibody or anti HBc antibody tests, and positive with HBV-DNA quantitative test
5. Pregnant, suspected pregnant, or lactating
6. Patients who have Psycosis or psychiatric symptoms are judged inappropriate for participation in the trial
7. Patients who need the treatment with continued use of flucytosine, phenytoin, or warfarin potassium
8. Patients who have a medical history of allergy to iodine
9. Patients who have hypersensitivity to docetaxel, cisplatin, and drug-containing polysorbate 80
10. Patients who have a complication or a history of highly sensitive reactions to antibody formulations
11. Even if insulin or oral hypoglycemic agent is continued use, the result of HbA1c test is 6.5% or more in JDS or 6.9% or more in NGSP
12. Patients who have advanced pulmonary emphysema, which is observed by pulmonary function test or CT test
13. Patients who have uncontrollable hypertension
14. Patients who have unstable angina or a medical history of myocardial infarction within 6 months before enrollment
15. Patients who have diverticulitis or symptomatic peptic ulcer disease
16. Patients who have a history of transplantation therapy, such as hematopoietic stem cell transplantation
17. Patients who have a medical history of treatment with an anti-PD-1 antibody, anti-PD-L1 antibody, anti-PD-L2 antibody, anti-CD137 antibody, anti-CTLA-4 antibody, or any other antibody for inhibition or modulation of T cell costimulatory pathway or cancer vaccine."

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2019-05-07 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Rate of participants with dose limiting toxicities (DLTs) | from initial dose to 30 post-operative days
  To evaluate the safety of combination chemotherapy with nivolumab as neoadjuvant Tx

SECONDARY OUTCOMES:
Response rate (RR): percentage of participants with with a best response of CR or PR | from baseline to date of disease progression, approximately 24 months
  To evaluate the efficacy of combination chemotherapy with nivolumab as neoadjuvant Tx
Pathological complete response rate | from baseline to operation, average of 10 weeks after initial dose
  To evaluate the efficacy of combination chemotherapy with nivolumab as neoadjuvant Tx
Radical resection rate | at operation, average of 10 weeks after initial dose
  To evaluate the efficacy of combination chemotherapy with nivolumab as neoadjuvant Tx
Treatment completion rate | from baseline to operation, average of 10 weeks after initial dose
  To evaluate the efficacy of combination chemotherapy with nivolumab as neoadjuvant Tx
Adverse event (AE) expression rate | up to 30 postoperative days
  To evaluate the safety of combination chemotherapy with nivolumab as neoadjuvant Tx
Progression-free survival (PFS) | from baseline to date of disease progression or death, approximately 24 month
  To evaluate the efficacy of combination chemotherapy with nivolumab as neoadjuvant Tx
Overall survival (OS) | from baseline to date of death, approximately 24 month
  To evaluate the efficacy of combination chemotherapy with nivolumab as neoadjuvant Tx

CONTACTS AND LOCATIONS:
Overall Officials: Ken Kato, MD/PhD, Study Chair — Department of Gastrointestinal Medical Oncology, National cancer center hospital
Locations (1):
- National Cancer Center Hospital, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yamamoto S, Kato K, Daiko H, Kojima T, Hara H, Abe T, Tsubosa Y, Nagashima K, Aoki K, Mizoguchi Y, Kitano S, Yachida S, Shiba S, Kitagawa Y. Feasibility study of nivolumab as neoadjuvant chemotherapy for locally esophageal carcinoma: FRONTiER (JCOG1804E). Future Oncol. 2020 Jul;16(19):1351-1357. doi: 10.2217/fon-2020-0189. Epub 2020 May 12. PMID 32396014